CLINICAL TRIAL: NCT02615444
Title: An Investigation of the Effects of Consuming Oatcakes Containing 4g of Oat Beta-glucan on Physiological Parameters in Individuals at Risk of Developing Metabolic Syndrome
Brief Title: The Effects of Beta-glucan Enriched Oatcake Consumption on Metabolic Disease Risk Factors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Queen Margaret University (Other)
Responsible Party: Principal Investigator, Suzanne Zaremba, PhD Student, Queen Margaret University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: QueenMUsz
Record Dates: First submitted 2015-11-05; First posted 2015-11-26 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Metabolic Syndrome X; Cardiovascular Diseases
Keywords: Metabolic Syndrome X; Overweight; Waist Circumference; Blood Pressure; Cholesterol; Oat beta glucan
MeSH Terms: conditions — Metabolic Syndrome; Cardiovascular Diseases; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beta-glucan enriched oatcake (Experimental): Oatcakes which have been enriched with beta-glucan. Each participant will consume 5 oatcakes daily in order to ingest 4g of oat-beta glucan.
  Interventions: Dietary Supplement: Beta-glucan enriched oatcake
- Isocaloric control (Placebo Comparator): Control: Wheat based snack, equicaloric and matched to intervention product for macronutrient content. Contains no oat-beta glucan. Each participant will consume 6.5 Krackawheats daily.
  Interventions: Dietary Supplement: Isocaloric control

INTERVENTIONS:
Dietary Supplement: Beta-glucan enriched oatcake — 5 oatcakes enriched with oat beta-glucan will be consumed daily for six weeks
  Arms: Beta-glucan enriched oatcake
Dietary Supplement: Isocaloric control — 6.5 wheat based control snacks without beta-glucan will be consumed daily for six weeks
  Arms: Isocaloric control

SUMMARY:
The purpose of this study is to determine whether daily consumption of soluble fibre, oat beta glucan (4g), for six weeks will have any impact on overweight/obese individuals in terms of risk factors used to define metabolic disease.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether daily consumption oat beta glucan (4g) for six weeks will have any impact on overweight/obese individuals in terms of risk factors used to define metabolic disease.

Oat beta-glucan has been incorporated into a novel oatcake product manufactured by Nairn's Oatcakes Ltd. Consumption of the oatcake products will deliver enough oat-beta glucan to the diet to meet European Food Safety Authority health claims for lowering blood cholesterol and reducing post-prandial glycaemic responses.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years and older
* Waist circumference measurements of ≥94cm for males and 80cm for females, or a body mass index of ≥30kg/m2
* Individuals who are able to provide informed consent

Exclusion Criteria:

* Postmenopausal females
* Smokers
* Individuals who suffer from, or taking medication for, cardiovascular or gastro-intestinal disease
* Impaired glucose tolerance/Diabetes mellitus
* Pregnancy or breastfeeding
* Those who have high dietary fibre intakes (>20g/day)
* Known food allergies to oats, wheat, lactose, or sesame seeds

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Waist Circumference | 6 weeks

SECONDARY OUTCOMES:
Blood Pressure | 6 Weeks
Fasting Serum Triglycerides | 6 weeks
Oral Glucose Tolerance Test | 6 weeks
Fasting Serum HDL Cholesterol | 6 Weeks
Fasting Serum total Cholesterol | 6 weeks
Interleukin-6 | 6 weeks
Energy Intakes (kilocalories) and Macronutrient intakes (grams) from food diaries | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Zaremba, Study Chair — Queen Margaret University
Locations (1):
- Queen Margaret University, Edinburgh, Musselburgh, East Lothain, United Kingdom

REFERENCES:
- [Background] Pouliot MC, Despres JP, Lemieux S, Moorjani S, Bouchard C, Tremblay A, Nadeau A, Lupien PJ. Waist circumference and abdominal sagittal diameter: best simple anthropometric indexes of abdominal visceral adipose tissue accumulation and related cardiovascular risk in men and women. Am J Cardiol. 1994 Mar 1;73(7):460-8. doi: 10.1016/0002-9149(94)90676-9. PMID 8141087
- [Background] Lissner L, Lindroos AK, Sjostrom L. Swedish obese subjects (SOS): an obesity intervention study with a nutritional perspective. Eur J Clin Nutr. 1998 May;52(5):316-22. doi: 10.1038/sj.ejcn.1600567. PMID 9630380
- [Background] Howarth NC, Saltzman E, Roberts SB. Dietary fiber and weight regulation. Nutr Rev. 2001 May;59(5):129-39. doi: 10.1111/j.1753-4887.2001.tb07001.x. PMID 11396693
- [Background] Liatis S, Tsapogas P, Chala E, Dimosthenopoulos C, Kyriakopoulos K, Kapantais E, Katsilambros N. The consumption of bread enriched with betaglucan reduces LDL-cholesterol and improves insulin resistance in patients with type 2 diabetes. Diabetes Metab. 2009 Apr;35(2):115-20. doi: 10.1016/j.diabet.2008.09.004. Epub 2009 Feb 20. PMID 19230737